CLINICAL TRIAL: NCT04011488
Title: Shared Decision Making and How it Impacts Patient Understanding: Using an Interactive Knee Osteoarthritis App Based on a Cost Model to Generate a Patient Shared Decision Making Tool: Multi-center Randomized Clinical Trial Study Protocol
Brief Title: Shared Decision Making and How It Impacts the Patient Understanding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient recruitment
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: University of Pennsylvania (Other); Johns Hopkins University (Other); 3rd Coast Research Associates (Unknown); Yale University (Other); University Hospitals Cleveland Medical Center (Other); PIH Family Practice Residency (Unknown); Baylor College of Medicine (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-462
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: shared decision making
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard patient information data sheet (No Intervention)
- SDM Tool (Experimental): A simple, one-page tool that provides a framework for the patient discussion, which improves the consistency of the patient-provider communication. This SDM can also be customized to a specific patient based on gender, race/ethnicity, age, and select comorbidities (obesity, hypertension and diabetes).
  Interventions: Other: Shared Decision Making Tool

INTERVENTIONS:
Other: Shared Decision Making Tool — We've used the framework from this model and adapted it to the patient perspective to create a Patient Shared Decision Making Tool. The model is interactive so it can be customized to a specific patient. It has adjustments built in for gender, race/ethnicity, age, and select comorbidities (obesity, hypertension and diabetes).
  The strongest, underlying message is that any treatment choice is better than not seeking treatment. To illustrate this, a "Do Nothing" pathway is included for comparison purposes.
  Arms: SDM Tool

SUMMARY:
Shared Decision Making (SDM) supports patient centered care and improves patient outcomes and satisfaction. Movement is Life (MIL) created an innovative SDM tool to provide a personalized framework for discussion of the projected impact to patients of their decisions regarding treatment options for knee osteoarthritis.

1. Did use of the MIL SDM tool for knee osteoarthritis result in an increased level of self-reported physical activity at one month in African American and Hispanic women?
2. Did use of the MIL SMD tool increase subject likeliness to recommend the physician?
3. What is the qualitative feedback from subjects on ease of use of the MIL SDM tool?

ELIGIBILITY:
Inclusion Criteria:

* - Aged 45 to 64 years
* Mild to moderate knee pain consistent with a diagnosis of osteoarthritis by the clinician
* Self-identified as African American and/or Hispanic
* At least one of the following comorbidities:

  1. Obesity (BMI ≥ 30),
  2. Hypertension (ICD10 codes below)
  3. Diabetes (ICD10 codes below)

Exclusion Criteria:

* - Known inflammatory arthritis (Lupus, Sjogrens, rheumatoid arthritis)
* Prior total knee replacement
* Recommended total knee replacement
* Acute knee trauma

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Survey | One month afterwards
  The primary outcome instrument is the Patient Information Survey administered shortly after the evaluation. There is both a qualitative and quantitative portion of the survey.

SECONDARY OUTCOMES:
Personal Health Questionnaire (PHQ-8), | One month post intervention
  Depression Survey
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS,JR) | One month post intervention
  joint specific functional outcome survey
Patient Experience Survey | One month post intervention
Patient Information Survey- Qualitative portion | One month post intervention
Shared Decision Making (SDM) Survey | One month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Parks, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Michael L. Parks, MD, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No